A Motivational Training Program for Secondary Physical Education Teachers Based on the Circumplex Model: A Study Protocol of a Randomized Controlled Trial.

#### Abstract

Introduction: In most Self-Determination Theory (SDT) research, improving (de)motivating teaching styles enables numerous benefits for students and teachers, although there is less evidence on the latter. Although the recent circumplex model provides a fine-grained picture of the different (de)motivating teaching styles (i.e., autonomy support, structure, control, and chaos) that physical education (PE) teachers can use in their lessons, no previous motivational training programs have been based on this model. Moreover, all SDT-training programs have been implemented through different group sessions, but individual sessions have not also been delivered.

**Objective**: This study outlines the protocol of a motivational training program, derived from the circumplex model, designed to enhance (de)motivating teaching styles among PE teachers. Consequently, this program seeks to improve motivational variables and influence (mal)adaptive outcomes in both teachers and students.

**Design**: A randomized controlled trial design with a mixed-method approach.

**Participants:** At least 16 secondary PE teachers will be assigned to either an experimental group or a control group, together with part of their students.

**Intervention**: The training program comprises four face-to-face group sessions and two follow-up sessions (one individual and one group sessions). PE teachers will learn how to support autonomy and provide structure, as well as to be less controlling and chaotic towards students. Over a period of approximately five months, teachers will implement these motivational strategies during their PE classes.

Outcome measures: Different (de)motivating teaching styles, motivational variables, and (mal)adaptive outcomes will be assessed in both PE teachers and their students at three distinct

points: before the training program (T1), during the intervention (T2) and at the end of the intervention (T3). Additionally, two discussion groups involving all experimental PE teachers will be held (one following the training program and another at the end of the intervention).

**Conclusion**: The results from this study could be useful for developing motivational training programs for in-service PE teachers.

Trial registration: (AÑADIR)

**Keywords:** circumplex approach, motivating styles, professional development, selfdetermination theory, psychological needs, motivation.

#### Introduction

Physical Education (PE) teachers hold a pivotal role in guiding students through their learning process. Drawing on Self-Determination Theory (SDT; Ryan & Deci, 2020), teachers' (de)motivating style, referred to as "the interpersonal sentiment and behaviour that teachers rely on during instruction to motivate students to engage in and benefit from learning activities" (Reeve et al., 2014, p. 94), is a crucial element in the teaching process. Recent research suggests that PE teachers employ a diverse array of teaching behaviours in their educational practice (Burgueño, García-González, et al., 2024). Autonomy, competence, and relatedness-supportive teaching behaviours (i.e., need-supportive teaching behaviours) have been positively related to students' autonomous motivation and adaptive outcomes in PE, while the opposite is true for autonomy, competence, and relatedness-thwarting behaviours (i.e. need-thwarting behaviours) (Vasconcellos et al., 2020; White et al., 2021). Consequently, continuous development teaching (CDT) programs, based on SDT (Ryan & Deci, 2017), has increased in the last years. These SDT-training programs, mainly focused on autonomysupportive strategies, revealed positive effects on students' perceptions of (de)motivating teaching behaviours and motivational outcomes (Vasconcellos et al., 2020). Over the past decade, SDT-training programs have also demonstrated positive effects on teachers' selfperceptions of certain antecedents, support for autonomy and structure, and various motivational and (mal)adaptive outcomes (Reeve & Cheon, 2021). However, additional research is required, as most studies have not focused on reducing need-thwarting behaviours.

Recently, grounded in SDT (Ryan & Deci, 2017), the circumplex model (Aelterman et al., 2019) offers a detailed view of the different (de)motivating teaching styles (i.e., autonomy support, structure, control, and chaos) that teachers can adopt in their classes. This circumplex model delineates eight teaching approaches across these four teaching styles (Aelterman et al., 2019; Escriva-Boulley et al., 2021). To develop the most effective

interventions, it is crucial for researchers to understand the effectiveness of motivational training programs, not only in terms of the four (de)motivating teaching styles but also across the eight specific teaching approaches. Yet, no existing motivational training programs have incorporated this new circumplex approach. This mixed-method study sets out to expand existing knowledge by describing a protocol for a motivational training program based on the circumplex model, aimed at enhancing (de)motivating teaching styles, as well as (mal)adaptive outcomes among PE teachers and their students.

# Self-Determination Theory: The Importance of Basic Psychological Needs in Teaching

According to SDT (Ryan & Deci, 2017), PE teachers need to satisfy the three basic psychological needs (i.e., autonomy, competence, and relatedness) in teaching to experience well-being and feel fulfilled in their job. However, it has been established that these needs can also be frustrated (Vansteenkiste et al., 2020). Autonomy satisfaction is linked with PE teachers' sense of making their own decisions and implementing their ideas in lessons, while autonomy frustration arises from feelings of compulsion to teach in prescribed ways and experiencing pressure in work-related tasks. Competence satisfaction involves PE teachers' perception of success and effectiveness in their PE lessons, whereas competence frustration refers to experiencing feelings of ineffectiveness and failure in their teaching-related tasks. Lastly, relatedness satisfaction is experienced by PE teachers when they feel connected and integrated with colleagues and students, while relatedness frustration occurs when they feel isolated and excluded in their work environment (Ryan & Deci, 2017; Vansteenkiste et al., 2020). According to SDT, teachers' need satisfaction and frustration can be influenced by several antecedents including contextual factors, personal factors, and perceptions of others' behaviours and motivation (Haerens et al., 2016; Matosic et al., 2016). Moreover, in alignment with SDT, these PE teachers' need-based experiences significantly influence their well-being and play a crucial role in the (de)motivating teaching styles they adopt during PE

lessons. Previous SDT-based research (Slemp et al., 2020), indicates that teachers' need satisfaction is positively associated with different adaptive outcomes (e.g., well-being, job satisfaction, engagement, etc.), and need-supportive teaching behaviours towards students. However, teachers' need frustration has been positively related to maladaptive outcomes (e.g., distress, burnout, etc.) and need-thwarting teaching behaviours towards students. Therefore, addressing certain antecedents of (de)motivating teaching styles could enhance teachers' need satisfaction and reduce their frustration, consequently facilitating the adoption of motivating teaching behaviours.

# A Fine-Grained Picture of (De)Motivating Teaching Styles: A Circumplex Model

The circumplex model offers a deeper and detailed perspective of the four teaching styles that a PE teacher can employ in his/her lessons (Aelterman et al., 2019). These styles are categorized along two axes: one horizontal, indicating whether the style supports or thwarts students' needs, and one vertical, reflecting the degree of the directiveness exhibited by the PE teachers. Each teaching style is further divided into two distinct approaches, culminating in a total of eight specific teaching approaches (Aelterman et al., 2019).

On the one hand, the first motivating teaching style, characterized by low directiveness and high need-supportive, is termed autonomy support. PE teachers who demonstrate a tone of receptivity and flexibility to accommodate the preferences and interests of their students provide an autonomy-supportive environment (Vansteenkiste et al., 2019). Autonomy support can emerge by a participative (i.e., PE teacher provides students with choices and decision-making power) and an attuning teaching approach (i.e., PE teacher fosters students' interests, accepts expressions of negative affect, and explains the relevance of each activity performed). The second motivating teaching style, characterized by high directiveness and high need-supportive, is termed structure (Aelterman et al., 2019). Structure involves PE teachers adopting attitudes oriented towards progress and process, always

considering the ability levels and the needs of each student (Vansteenkiste et al., 2019). The structuring style is displayed by a guiding (i.e., PE teacher provides students with helpful guidelines and encouragement for successful task completion) and a clarifying teaching approach (i.e., PE teacher communicates the goals and expectations of the lessons to the students) (Escriva-Boulley et al., 2021).

On the other hand, the first demotivating teaching style, characterized by high directiveness and high levels of need-thwarting, is termed control. It refers to those PE teachers who exert pressure on students to think, feel, and behave in specific ways (Vansteenkiste et al., 2019). This controlling style can be expressed by a demanding (i.e., PE teacher imposes mandatory actions on their students and administer punishment or threats if they fail to comply) and a domineering teaching approach (i.e., PE teacher uses manipulative strategies such as inducing shame, disapproval, or even humiliation to comply with their requests) (Burgueño, Abós, et al., 2024). The second demotivating teaching style, characterized by low directiveness and high levels of need-thwarting, is termed chaos. It refers to those PE teachers who adopt a laissez-faire approach, characterized by their unpredictable and inconsistent behaviour (Vansteenkiste et al., 2019). Chaotic style is expressed by an abandoning (i.e., after multiple failed attempts, the PE teacher resigns and leaves the students to fend for themselves) and an awaiting teaching approach (i.e., PE teachers do not plan lessons extensively as they prefer to wait and see how things unfold) (Aelterman et al., 2019).

Previous studies based on SDT and the circumplex model (Burgueño, Abós, et al., 2024; García-Cazorla et al., 2024) have shown that teachers who have their needs satisfied implement autonomy-supportive (i.e., participative and attuning approaches) and structuring styles (i.e., guiding and clarifying approaches) in their PE, while those teachers who have their needs frustrated, use controlling (i.e., demanding and domineering approaches) and

chaotic styles (i.e., abandoning and awaiting approaches). According to SDT, the adoption of these (de)motivating teaching styles/approaches by PE teachers may elicit various motivational consequences for students.

# Influence of (De)Motivating Teaching Approaches on Students' Motivational Outcomes

Grounded in the circumplex model, a growing body of research examines the relationship between (de)motivating teaching styles/approaches and students' motivational outcomes. For example, Burgueño, Abós, et al. (2024) demonstrated that students' perceptions of autonomy-supportive (i.e., participative and attuning) and structuring (i.e., guiding and clarifying) styles from PE teachers are positively related to students' needs satisfaction, but also the clarifying approach is negatively associated with students' need frustration. Diloy-Peña et al. (2024) also showed that those students who perceived autonomy-supportive and structuring styles and approaches reported higher values in positive PE experiences, learning in PE, and intention to participate in physical activity (PA). Conversely, Burgueño, Abós, et al. (2024) showed that controlling (i.e., demanding and domineering approaches) and chaotic (i.e., abandoning and awaiting approaches) styles are positively associated with students' needs frustration, but also the domineering and abandoning approaches are negatively associated with students' need satisfaction. Additionally, comprehensive SDT-based research in PE indicates that students' need satisfaction is positively related to autonomous motivation and positive behavioral, affective, and cognitive outcomes, while students' need frustration is positively related to controlled motivation, amotivation, and various maladaptive outcomes (Vasconcellos et al., 2020). Consequently, given the associated benefits for students, SDT-training programs aimed at improving PE teachers' motivating teaching syle have increased in recent years.

Previous SDT-Training Programs for PE Teachers and Added Value of this Study.

SDT-training programs have predominantly concentrated on autonomy-supportive strategies, revealing positive effects on students' perceptions of their PE teachers' (de)motivating teaching styles/approaches, as well as on motivational outcomes in PE lessons (Vasconcellos et al., 2020). A previous review of SDT-training programs also suggested that PE teachers can benefit from participating in these programs, although more research is needed to examine their effects on a wide range of outcomes (Reeve & Cheon, 2021). However, there are very few SDT-training programs that examine their effects on both students and teachers. For example, Cheon et al. (2020), showed that PE teachers who participated in an eight-hour, three-session face-to-face SDT-training program, focused on provided structure in an autonomy-supportive way, showed improvements across all assessed variables (i.e., teacher-reported autonomy support and structure, teaching efficacy, intrinsic instructional goals, harmonious passion, job satisfaction, and relationship satisfaction with students). Moreover, students also perceived improvements in autonomy and structure support, autonomy and competence satisfaction, and outcomes such as classroom engagement, skill development, anticipated PE performance, and future intention to do PA. It is noteworthy that in most of these SDT training programs, the effects on teachers have only been assessed after they implemented the strategies with the students (Aelterman et al., 2013). Gaining insight into teachers' perspectives both before the training, immediately after the SDT-training program, and upon completion of the entire intervention, could also enhance the acceptance, sustainability, and scalability of the program. To achieve this, employing a qualitative methodology could build on existing findings, providing greater justification for the results obtained (in addition to quantitative).

To the best of our knowledge, no previous motivational training programs have been designed based on the circumplex model. This model can guide the teaching approaches associated with each of the (de)motivating styles and provide a better understanding of the

potential effects of the program on each of the eight teaching approaches. In the educational domain, only three programs to date have examined the effects of SDT-training programs on (de)motivating teaching styles using the Situations-in-School Questionnaire (SIS; an instrument to assess the eight teaching approaches proposed by the circumplex model) (Cheon et al., 2020; Conesa et al., 2023; Jang et al., 2023). However, none of these programs have specifically examined the effects of all the eight teaching approaches proposed by the circumplex model. In addition, few SDT-training programs have focused on reducing controlling and chaotic teaching styles. Since teachers may combine need-supportive and need-thwarting approaches (Burgueño, García-González, et al., 2024), it seems necessary for these programs to also focus on reducing these behaviors.

The characteristics, content, and implementation mode of the SDT-training programs also appear to be crucial factors to consider. To date, all SDT-training programs have been implemented through different group sessions with PE teachers. However, different person-centered studies have indicated that each PE teacher may exhibit a very different (de)motivating teaching style profile (Burgueño, García-González, et al., 2024). For instance, one teacher might employ both autonomy-supportive and structuring styles, alongside a controlling style. Conversely, another teacher might use autonomy-supportive behaviours while lacking structure, resulting in a chaotic classroom environment. Therefore, it seems necessary that at least part of the motivational training program be individualized to the (de)motivating teaching profile and personal characteristics of each teacher. The use of observational methodology in teacher' own classes has emerged in recent years as a solution to provide constructive and individual feedback through videos (Bouten et al., 2023). However, to date, it has only been used in SDT-training programs to examine intervention fidelity and/or to assess possible changes in the (de)motivating teaching styles (Reeve & Cheon, 2021). Combining a brief initial theoretical component with a more extensive

practical part (i.e., microteaching) has been previously identified as essential for applying what has been learned in contexts as close to reality as possible (Aelterman et al., 2013). Ultimately, the adoption of a congruent style, where trainers implement the program using (de)motivating teaching styles has also been positively perceived by PE teachers. This approach allows them to observe real-life examples of how to implement these strategies effectively (Aelterman et al., 2013). Moreover, in line with SDT, it could lead to an immediate effect on the teachers' need satisfaction during the training that has been positively associated with effectiveness and feasibility beliefs in terms of autonomy support and structure, as well as teachers' intentions to apply the proposed strategies (Aelterman et al., 2016).

Finally, while previous studies have considered gender as a covariate to analyze the effects of SDT-based interventions, gender differences in study variables are seldom reported for both teachers and students. Given prior SDT-related research indicating that (de)motivating teaching behaviours may be perceived differently by boys and girls students (White et al., 2021) and male and female teachers (García-Cazorla et al., 2024), it is crucial to determine whether the intervention is equally effective for both genders to mitigate any potential gender-related inequities.

To extend previous knowledge, this mixed-method study describes the protocol of a motivational training program, based on the circumplex model, aimed at improving (de)motivating teaching styles/approaches among PE teachers. The first hypothesis suggests that the features of the motivational training program will be positively perceived by PE teachers (H1). We also hypothesize that experimental school female and male teachers will perceive improvements in several antecedents, autonomy and competence satisfaction/frustration at work, (de)motivating teaching styles/approaches, and (mal)adaptive outcomes at least at the end of the intervention implementation toward students (H2). Finally,

both boys and girls from experimental groups will perceive improvements in their PE teachers' (de)motivating teaching styles/approaches, autonomy and competence satisfaction/frustration in PE, and adaptive outcomes in PE lessons (H3).

### Materials and methods

## Context, design, and randomization

This study will be carried out in a northeast region of Spain [details masked for review process]. PE is mandatory for every secondary school student in Spain. Each student receives two 50-minute coeducational PE lessons per week. Spanish Secondary PE teachers are expected to teach between 18 and 21 hours per week. Typically, the annual teaching plan of PE teachers includes approximately six to eight distinct teaching units per year. These units encompass various content types such as individual, cooperative, and interactive sports and games, as well as body expression, health-related fitness, and outdoor activities, all of which are outlined in the PE curriculum. The academic year lasts from September to June, divided into three terms, each separated by a holiday period (i.e., Christmas and Easter).

A randomized controlled trial design with a mixed-method approach will be carried out. PE teachers agreeing to participate in the trial will be randomly assigned to either the experimental or the control group. Randomization will be conducted using the digital tool available at <a href="https://echaloasuerte.com/">https://echaloasuerte.com/</a>. To prevent contamination of the experimental condition, schools will only participate in one group (i.e., experimental or control). Subsequently, at least two groups of students from each PE teacher will be randomly selected.

This study will comprise two phases: 1) a teacher-training phase and 2) an implementation phase with students. It should be noted that the training program will continue with some individual and group sessions during the implementation phase. Since teachers' and students' perceptions of (de)motivating teaching styles and approaches and other study variables require several months for greater accuracy in their perceptions, the

training program will not start until the second term of the academic year (for more details see Figure 1).

Figure 1. Characteristics of the training program and timeline for data collection



**Notes**: \*the variables assessed in PE teachers and students are detailed in the corresponding section; \*\*the training program has two follow-up sessions (individual and group).

The study has been approved by the Ethics Committee of the University of [details masked for review process] and follows all ethical procedures established in the Declaration of Helsinki.

#### Sample size calculation

The sample size for this intervention-based study was calculated using R Studio to ensure adequate power in the detection of potential statistically significant effects.

Considering a multi-level design nesting center, PE teacher and group, the sample size calculation was grounded on an anticipated effect size of 0.5, reflecting a moderate impact of the intervention. The power of the study was set at 80% with a significance level (alpha) of 0.05, aligning with common practices in educational research (McConnell et al., 2019).

Acknowledging the inherent structure of this study, an Intra-Class Correlation (ICC) of 0.1 was assumed based on similar educational settings (Hedges & Hedberg, 2007). This ICC estimate accounted for the expected homogeneity within the three levels (class group within PE teacher, PE teacher within center). To accommodate potential participant dropout, particularly among students, we incorporated a 40% anticipated dropout rate into our calculations (e.g., Meerits et al., 2022). The minimum sample size was adjusted to 210 students across 15 PE teachers, averaging 14 students per teacher. This adjustment ensures that our study maintains sufficient statistical power even in the face of anticipated losses, thereby safeguarding the integrity and validity of our findings.

## Participants and recruitment

At least 16 secondary PE teachers, eight in the experimental group and eight in the control group, along with their respective students, will be expected to participate in this study. The maximum number of participating teachers will be capped at 20, due to the limited human resources of the research team. PE teachers will select at least two classroom groups comprising at least 14 students each to invite to participate in this study. Eligible students will be those aged 12 to 17 years in secondary schools. Participation will be voluntary and anonymous.

Various social media platforms (i.e., Instagram, Twitter, and WhatsApp) and other communication methods (i.e., email) will be used for teachers' recruitment. An informative poster will be launched, detailing the target sample, content, aims, and training program dates. This poster will also include two links (QR code): one with a document providing further information and another to registration through a brief Google Forms questionnaire. Regarding the additional information document, it is important to note that it will detail a more comprehensive overview of the objectives, the different phases of the program, inclusion criteria, the requirements that each teacher must accept to participate, and the

teaching skills that will be developed during the training program. Teachers with further inquiries can contact the research team via email or phone. The registration period will last approximately 21 days.

Once the interested PE teachers have registered, various inclusion criteria will be considered for the final selection: 1) Being an in-service PE secondary school teacher for the entire academic year; 2) Attending 100% of the training program sessions; 3) Fill in a short questionnaire at the end of each session of the training program, as well as fulfilling questionnaires of the study variables three times; 4) Allowing the recording of two PE lessons; 5) Participating in two focus groups, one at the end of the training program and one at the end of the study, and 6) Not participating in other training sessions related to PE instruction during the program. Moreover, the inclusion criteria for students will be: 1) Authorization from parents or legal guardians; 2) Completion of questionnaires of the study variables three times; 3) Regular participation in PE lessons.

## Measures

# **Questionnaires**

The following PE teachers' variables will be measured using Google Forms before the training program (T1), as well as during (T2) and at the end of the implementation of the intervention with their students (T3) (see Figure 1):

**Socio-demographic variables**. Age, gender, teaching experience, type of school (public or private), and school location (rural or urban) will be self-reported by teachers.

(De)motivating teaching styles and approaches towards students. To assess self-reported (de)motivating teaching styles toward students, the Spanish version of the SIS in Physical Education (SIS-PE; (Burgueño, Abós, et al., 2024) will be used. The SIS-PE comprises 12 typical teaching situations consisting of four items each (i.e., 48 items).

Autonomy-supportive items are categorised into participative (four items) and attuning (eight

items) approaches. Structure items are operationalised into guiding (seven items) and clarifying (five items) approaches. Control items are divided into demanding (seven items) and domineering (five items) approaches. Chaos items are operationalised into abandoning (eight items) and awaiting (four items) approaches. For instance, this situation "At the start of class..." is followed by four items: you can explore students' prior knowledge of the topic (attuning), set up a class clearly and straightforwardly (clarifying), demand application of what's taught (demanding), or just begin and let the class evolve (awaiting)". It should be noted that, since teachers' perceptions of their (de)motivating teaching styles could be different according to the classroom group, teachers will have to answer the questionnaire taking into account the groups of students selected for the study. Teachers' responses will be assessed using a 7-point Likert scale ranging from 1 ("Does not describe me at all") to 7 ("Describes me perfectly").

Autonomy and competence satisfaction and frustration at work. To assess PE teachers' perceptions of autonomy and competence satisfaction and frustration at work, the Spanish version of the Basic Psychological Needs at Work Scale for in-service teachers (Abós Catalán et al., 2018) and the Basic Psychological Need Satisfaction and Frustration Scale (Chen et al., 2015), will be used, respectively. Four of the six factors of these scales will be assessed, except relatedness satisfaction and frustration. Both scales are preceded by the stem "In my job as a PE teacher..." assessing autonomy satisfaction (Four items; e.g., "My job allows me to make decisions"), autonomy frustration (Four items; e.g., "I feel that most of the things I do in my job, I do them because I have to do them"), competence satisfaction (Four items; e.g., "I have the ability to do my job well"), and competence frustration (Four items; e.g., "I have serious doubts that I can do well in my job"). Teachers' responses will be assessed using a 5-point Likert scale ranging from 1 ("strongly disagree") to 5 ("strongly agree").

**Job satisfaction at work.** Teachers' perceptions of job satisfaction at work will be assessed using a Spanish translation (Abós et al., 2019) of the Teacher Job Satisfaction Scale (TJSS; Skaalvik & Skaalvik, 2011). This four-item scale includes one single factor (e.g. "I enjoy working as a teacher"). Teachers' responses will be registered on a 6-point Likert scale from 1 ("strongly disagree") to 6 ("strongly agree").

Emotional exhaustion at work. Teachers' emotional exhaustion will be assessed using the Spanish version of the Maslach Burnout Inventory-General Survey (Gil-Monte, 2002). In line with other studies on PE teachers (Richards et al., 2019), only the five items assessing the exhaustion factor will be used in the present study (e.g., "I feel burned out from my work"). Teachers' responses will be reported on a 7-point Likert scale from 0 ("never") to 6 ("every day").

**Job performance.** Teachers' perceptions of their professional performance will be assessed using the following sentence: "Rate your satisfaction with your professional performance this academic year", which has been previously used in other studies (Barrick et al., 2002). Teachers' responses will be provided on a 9-point Likert scale, ranging from 1 ("non-existent") to 9 ("excellent").

Quality of the training program. Consistent with previous studies (Aelterman et al., 2013; Cheon & Reeve, 2015; Slingerland et al., 2017), a short paper-and-pencil questionnaire will also be measured immediately after each session of the training program carried out to gain insight into their content. Questions will be related to: (1) Interaction, (2) innovation, (3) interest, (4) intelligibility, (5) essentiality, (6) practical usefulness, (7) feasibility of the motivating strategies, (8) intention to implement the motivating strategies, (9) the extent to which one would recommend the training to others, (10) perceived changes in their (de)motivating styles, and (11) overall satisfaction. This questionnaire will be rated on a 5-point Likert scale from 1 (totally disagree) to 5 (totally agree), except for the last question, in

which teachers will rate the overall satisfaction on a scale from 1 to 10. Lastly, in an openended question, teachers will be able to detail the strengths and areas for improvement in each of the sessions to make slight adjustments to the training program in their future implementation.

Like their teachers, students will fill out the following questionnaires before the training program (T1), as well as during (T2) and at the end of the implementation of the intervention by the PE teachers (T3) (See Figure 1). Depending on the protocol of each school, these questionnaires will be completed in paper-and-pencil format or using Google Forms in a quiet classroom environment. The PE teacher will not be present when their students complete the questionnaires to avoid bias in the responses. In this sense, a member of the research will help the students with any doubts that may exist.

**Socio-demographic variables**. Age, gender, and school grade level will be self-reported by students.

(De)motivating teaching styles and approaches. To assess students' perceptions of (de)motivating teaching approaches of their PE teachers, the Spanish version of students of the Situations-in-School Questionnaire in Physical Education (SIS-PE; (Burgueño, Abós, et al., 2024) will be used. The only change in the instrument compared to the teachers' instrument is the structure of the sentences, as they are written from the students' perspective (e.g., "Your teacher invites you to suggest a set of norms or rules").

Autonomy and competence satisfaction and frustration in PE. To assess students' perceptions of autonomy and competence satisfaction in PE, the Spanish version (Zamarripa et al., 2020) of the Basic Psychological Need Satisfaction and Frustration Scale (Chen et al., 2015) will be used. Four of the six factors of these scales will be assessed, except relatedness satisfaction and frustration in PE. Preceded by the stem "In mi PE lessons...", the 16 items (four items per factor) assessing autonomy satisfaction (e.g., "I feel I have been doing what

interests me"), autonomy frustration (e.g., "I feel pressured to do too many tasks"), competence satisfaction (e.g., "I feel I can complete difficult tasks"), and competence frustration (e.g., "I feel like a failure because of the mistakes I make"). Items will be assessed using a 5-point Likert scale ranging from 1 (strongly disagree) to 5 (strongly agree).

**PE experiences.** In line with previous research (Diloy-Peña et al., 2024), students' perceived experiences in PE classes will be assessed using the question: "What are your experiences in PE lessons like?" The response possibilities were: (1) "very bad", (2) "bad", (3) "neutral", (4) "good", and (5) "very good".

**Perceived learning in PE.** In line with previous research (Diloy-Peña et al., 2024), students' perceptions of learning in PE will be assessed using the question: "How much do you learn in PE?" The response possibilities will be on a scale from 1 ("nothing") to 5 ("a lot").

Intention to be physically active. Students' perceptions of intention to participate in PA will be assessed using three items (e.g. "I intend to do active sports and/or physical activities during my leisure time in the next 5 weeks...") of the Spanish version of the Theory of Planned Behaviour Questionnaire (Tirado-González et al., 2012). This is a 5-point Likert scale from 1 ("strongly agree") to 7 ("strongly disagree").

# **Observation**

Observed (de)motivating teaching styles and approaches. Before the study, two raters with expertise in PE teaching instruction and the circumplex model will be trained in how to code (de)motivating teaching styles and approaches during PE using a Spanish translation of the SIS-PE-Coder, a new observation instrument that showed good reliability and internal validity (Van Doren et al., 2023). Following Van Doren et al. (2023) procedure, two randomly selected five-minute videos will be coded, trying to represent the beginning, middle or end of the lesson during six meetings. Before the final meeting, each expert

independently will code an entire lesson. Interobserver reliability was determined through Cohen's Kappa, using the following formula: agreements / (agreements + disagreements) × 100.

Consistent with the teachers' version of the SIS-PE, the SIS-PE-Coder consists of 41 items of which four items represent the participative approach, five items the attuning approach, six items the guiding approach, five items the clarifying approach, five items the demanding approach, seven items the domineering approach, five items the abandoning approach, and five items the awaiting approach. The coder will be prompted to assess each teaching behaviour from students' perspective, as specified by the statement: "If you were a student in this PE class, you would believe that the PE teacher...". Each item will be coded on a 7-point Likert scale, ranging from 0 (does not display this behaviour) to 6 (perfectly displays this behaviour). Two classes per experimental group teacher will be recorded by these two raters at two different moments of the implementation phase (before the second and third quantitative measures; See Figure 1). Items will be coded at 5-minute intervals (Aelterman et al., 2013). For every lesson, interval scores will be added together to create a sum score for each teaching behaviour throughout the entire duration of the lesson. This sum will be divided by the number of coded 5-minute intervals. Subsequently, scores for (de)motivating teaching styles, as well as the eight approaches, will be generated by averaging the scores of the individual items corresponding to each of the four styles and eight teaching approaches. The aim of the recordings will be not only to assess the fidelity of the intervention but also to provide opportunities for teachers to self-assessment, as well as coassessment by a member of the study.

For the observational analysis recordings, various professional video cameras will be used, as well as microphones connected to both the camera and the PE teacher who will be

conducting the lessons. For digitizing the video from the start to the end of the PE class, the iMovie (IOS) program will be used.

### Focus groups

Two discussion groups with all PE teachers will be held throughout the study (See Figure 1). Firstly, one focus group will be done immediately after the end of the fourth session of the training program. The main themes covered in the focus groups will be (1) the content of each session of the program (i.e., theoretical background, design of motivational strategies in different teaching units, and implementation of different PE lessons), (2) the didactical approach (e.g., images, videos, practical examples, formative assessment, and interactive exercises) and their perception of (de)motivating teaching style from de trainers (i.e., congruent teaching), (3) perceived changes in beliefs about (de)motivating teachers styles, the satisfaction of their basic psychological needs, and (de)motivating teaching styles towards students, and (4) overall assessment of the training (e.g., innovation, practical usefulness, feasibility of the motivating strategies, intention to implement the motivating strategies, satisfaction, etc.). This last question will complement the short questionnaire completed by the PE teachers at the end of each training program session (see above).

The second focus group will take place at the end of the intervention, coinciding with the completion of the teachers' and students' questionnaires in the post-test (T3). This will make it possible to find out the teachers' perception of the implementation phase, as well as of the different study variables. The main themes covered in the focus groups will be (1) the follow-up of the training program (e.g., individual and group sessions), (2) perceived changes in beliefs about (de)motivating teachers' styles, satisfaction of their basic psychological needs, (de)motivating teaching styles towards students, and job satisfaction, emotional exhaustion, and job performance.

Both focus group will be facilitated by a female with expertise in PE teaching instruction, the SDT framework, and qualitative methodology. To encourage open communication among PE teachers, the trainers will not be present during the group discussions. Focus group sessions will be started with an overview of both the aim and the procedure. The moderator will be supported by a co-moderator, tasked with managing logistics, recording notes, and overseeing the recording equipment. Furthermore, to conclude the focus group, the co-moderator will provide a summary of the primary viewpoints and will ask PE teachers whether these perceptions accurately reflect their views or if they wish to contribute additional insights.

Focus groups will take place in an empty, comfortable, and neutral room, lasting approximately 50 minutes. All sessions will be videotaped and transcribed to draw conclusions from the discussions.

# Teachers' Training Program and Intervention Implementation Towards Students

The intervention will comprise two phases in the experimental group: 1) a teacher-training phase (four face-to-face sessions and two follow-up sessions) and 2) an implementation phase where teachers will implement the strategies to the students (see Figure 1).

# Teachers' Training Program in the Experimental Group

The first part of the training program will last four weeks and eight hours in total. All PE teachers will participate in four weekly face-to-face group sessions, each two hours long, scheduled from 17:00 to 19:00. Grounded in the circumplex model, the sessions will aim to increase autonomy support and structure, while reducing controlling and chaotic approaches towards students. The training will be delivered by two members of the research team experienced in SDT-training programs for PE teachers.

The program incorporates strategies from established SDT-based teacher training programs (Aelterman et al., 2013; Cheon et al., 2020; Reeve et al., 2022; Reeve & Cheon, 2021). For example, to lead by example (i.e., congruent teaching), trainers provided autonomy support and structure and avoided control and chaos during all sessions of the training program. It is worth noting that the pre-test values on teachers' and students' perceptions of teaching approaches will allow the design of the training program to be individualized to the needs of the participants, particularly in the individual follow-up session.

The first two-hour face-to-face training session will unfold in a hybrid theoreticalpractical workshop format. It will commence with an introductory presentation by the trainers, followed by a brief review of the objectives and contents of the training program. The session will then transition into an autonomy-supportive exercise, where PE teachers will select a "getting-to-know-you" activity (15 min). Teachers should individually identify on a green sticky note some teaching behaviours of a good PE teacher they have had (e.g., "he/she allowed us to choose some tasks") and on a red sheet those of a bad PE teacher (e.g., "he/she constantly punished us"). Afterwards, once these sticky notes have been stuck on the board, teachers will have the opportunity to read and explain their experiences to the rest of the group (15 min). This activity will be linked to the theoretical background (i.e., SDT and circumplex model) that will be used throughout this training program. Thus, through ongoing collaboration and involvement of PE teachers (e.g., "What do you think the need for competence refers to?"), a concise overview of the SDT framework and circumplex model will be provided. This will be done using real-life examples and personal anecdotes shared by both the trainers and the teachers themselves (30 min). Finally, teachers will be encouraged to individually design a series of generic strategies to support autonomy and

provide structure, as well as to be less controlling and chaotic towards students in PE lessons (15 min). They will share these strategies with another teacher (15 min) and, finally, in pairs, with the entire group and trainers. This will lead to a collective reflection on the strategies themselves (e.g., "Why do you think this strategy might satisfy the need for autonomy?", "Could it satisfy or frustrate some other basic psychological need?") (25 min). At the end of the session, a brief explanation of the next steps and the objectives for upcoming sessions will be given to foster a positive disposition among the teachers. They will also be asked about the teaching units in their annual teaching plans that they still have to teach in each of the classroom groups involved in the study (5 min).

The second two-hour face-to-face training session will involve the design of motivational strategies in a practical workshop. In the first part of this session, a brief review of the previous session will be made, recalling theoretical background, identifying (de)motivating teaching behaviours, and reviewing the implementation in their PE lessons of the strategies proposed by PE teachers in the last session. For this, teachers will actively engage in the explanation process to assess the acquired learning (15 min). Afterwards, some videos of (de)motivating teaching strategies implemented by other secondary PE teachers will be shown. The videos will be selected based on teaching behaviours that have not been detailed by PE teachers in the previous training session (e.g., autonomy support; "provide an explanatory rationale"). Teachers will need to identify (de)motivating teaching behaviours depicted in the videos and consider their potential consequences on students' basic psychological needs satisfaction or frustration (25 min). Subsequently, the teaching units mentioned by the PE teachers in the previous training session will be listed. At least two of these teaching units will be chosen among all of them to design motivational strategies for small working groups (30 min). A coordinator of each group will present the different (de)motivating teaching strategies of the teaching unit and trainers and the rest of the teachers

will conduct a formative assessment of the co-created strategies (30 min). Finally, one teacher from each group will be offered the opportunity to teach one of the lessons of these teaching units to his/her colleagues, integrating at least two strategies from each (de)motivating teaching behaviour. The other teachers in the group will undertake to assist the volunteer teacher in designing the class.

The third two-hour face-to-face training session will involve applying and receiving the strategies learned throughout the training program in a simulated real-life situation (i.e., PE lesson) with the other participating teachers and other volunteers. One teacher from each group will teach one of the lessons of these teaching units using (de)motivating teaching behaviours (45 min per teacher). Afterwards, the trainers and the other PE teachers provided a formative assessment of positive strengths and areas for improvement (15 min after each class). Finally, another teacher will be encouraged to implement a lesson from the teaching unit of his or her annual teaching plan, with the help of the research team via Google Meet, in the last session of the training program.

The fourth face-to-face training session will focus on continuing the practical application of (de)motivating teaching strategies in a simulated real-life situation. This last session will be intended to be an example for the rest of the teachers in which a wide variety of (de)motivating teaching strategies appeared frequently. This last session will follow the same procedure as the previous class (45 min of class and 15 min of reflection). In the second part of the class, a final in-depth reflection on the first part of the training program will take place, focusing on synthesizing all the key concepts covered in the initial phase of the training program across the four sessions. Finally, teachers will receive a dossier of (de)motivating teaching behaviours organized in styles and approaches in line with the motivational behaviour change techniques (MBCTs) identified by themselves and the trainers in the training (see in the section on intervention implementation). Finally, the possibility of

creating a WhatsApp group will be offered to facilitate the follow-up of the training program.

Teachers will be able to share their progress, ask questions about the implementation of strategies, etc.

During the implementation phase, there will be one individual and one group followup sessions of the training program (see Figure 1) to monitor the implementation of strategies, give feedback on positive aspects and areas for improvement, and identify potential barriers or challenges encountered in the implementation of motivational strategies during this period. For the first follow-up session, the individual one, the trainers will visit each school to observe one PE class by each teacher. Subsequently, a detailed report of their teaching performance will be provided. The report will include: 1) a series of motivational strategies that the teacher used in their class, 2) a proposal of motivational strategies that the teacher could have used in their class, 3) a report of their teaching profile based on the pretest questionnaire values, including both the teachers' self-perception and the students' perceptions, and 4) advice and motivational strategies to improve their teaching profile in that specific class. For the second follow-up session, the group session, the objective will be to analyze the videos (taken from the first observational measure) of each teacher. The trainers will thoroughly review each video to extract clips showing each teacher using motivating and/or demotivating strategies. After each strategy is presented, a brief discussion will be held with the other teachers to identify strengths and possible improvement suggestions for these strategies. These follow-up sessions will be individualized and adapted to the needs of each teacher.

**Table 1**. Summary of the program training sessions.

| Face-to-face session 1 | Face-to-face session 2 | Face-to-face session 3 | Face-to-face session 4 | Follow-up<br>session 1 | Follow-up<br>session 2 |
|---|---|---|---|---|---|
| The entire | The entire | The entire | The entire | Individual | The entire |
| group of PE | group of PE | group of PE | group of PE | | group of PE |
| teachers | teachers | teachers | teachers | | teachers |

| 1. Presentation | 1. Summary of | <ol> <li>Application</li> </ol> | 1. Application | 1. Observation | 1. Observation |
|---|---|---|---|---|---|
| and getting-to- | the previous | of the | of the | of the PE | of the PE |
| know-you | lesson | motivational | motivational | teachers' real | teachers' real |
| activity | <ol><li>Identifying</li></ol> | strategies in | strategies in | classes and | classes and |
| <ol><li>Teaching</li></ol> | (de)motivating | two PE lessons | one PE lesson | subsequent | subsequent |
| behaviours of | teaching | of a simulated | of a simulated | constructive | constructive |
| good/bad | behaviours with | real-life | real-life | feedback. | feedback. |
| teachers. | real videos. | situation and | situation and | | |
| 3. Explanation | 3. Design of | subsequent | subsequent | | |
| of the | specific | reflection. | reflection. | | |
| theoretical | motivational | | 2. Summary of | | |
| backgrounds. | strategies in | | the key points | | |
| 4. Design of | different | | of the four | | |
| motivational | teaching units | | previous | | |
| strategies in PE | _ | | sessions | | |
| lessons. | | | | | |

# **Intervention Implementation Towards Students in the Experimental Group**

It should be noted that, although teachers will begin to apply some of the (de)motivating teaching styles and approaches from the first day they attend the training program, they will be implemented with greater variety, frequency, and intensity after the first part of the training (first four face-to-face sessions). The implementation phase will therefore last approximately five months, from January to the end of May. The training program that will be received by PE teachers will be focused on the motivational strategies proposed by Ahmadi et al. (2023). Teachers will be encouraged to implement as many MBCTs as possible in variety, frequency, and intensity in each of their PE classes.

# **Control group**

Control group teachers will not initially receive the training program and, as a result, will not intentionally implement any motivational strategy. They will only complete the questionnaires at the same times as experimental group teachers (See Figure 1). Control group teachers will receive the training program after the last study measurement, as well as an extensive final report on their teaching profile, and a series of motivational strategies aimed at enhancing their (de)motivating teaching style.

## Analysis plan

# Quantitative analyses

Firstly, the effects of the four sessions of the training program on the study variables assessed in teachers will be examined. The overall mean for each of the 11 variables perceived by PE teachers about the quality of the training program (e.g., interaction, innovation, interest, intelligibility, etc.) will also be calculated, representing the mean across the different sessions. A repeated measures analyses of variance (ANOVA) will be used to assess PE teachers' global appreciation of 11 variables related to the quality of the training program (e.g., interaction, innovation, interest, intelligibility, etc.) across the sessions of the training (i.e. within-subject analyses). Accordingly, each of the training sessions will be introduced as an independent variable (i.e. within-subject factor) and repeated measures of the PE teachers-related variables will be entered sequentially as dependent variables.

Secondly, the effects of the intervention implementation in PE lessons on study variables for both teachers and students will also be examined. Levene and Kolmogorov–Smirnov tests will be used to ensure the equality of variances and normal data distribution, respectively (p > .05). Cronbach's coefficient will be calculated for each study variable across the three measurements. To examine the effects of the intervention on study variables, a 3 x 2 (time x condition) repeated measures multivariate analysis of covariance (MANCOVA) will be performed for both teachers and students. Age, gender, teaching experience, type of school (public or private), and school location (rural or urban) will be introduced as covariates among teachers, while age, gender, and school grade level will be introduced as covariates among students. Subsequently, to examine intragender differences of the intervention on study variables, a 3 x 2 x 2 (time x condition x gender) repeated measures MANCOVA will be performed for both teachers and students. The same covariates will be entered as previously analysis, excluding gender. Multiple paired t-tests with Bonferroni correction will be calculated to determine between-group (i.e., experimental-control group) and within-group (i.e., pre-post) differences. Cohen's criteria will be used as indicators of small (.01), moderate

(.06), and large (.14) effect sizes (Field, 2017). All statistical analyses will be conducted using IBM SPSS Statistics v.25.0. Finally, a longitudinal structural equation model will be used to analyze the predictive relationships between the study variables, allowing for observation of potential differences at the three specific times (i.e., pre-test, middle, and post-test) when data are collected.

### Qualitative analyses

With respect to the qualitative data, both focus groups will be transcribed and analysed using NVivo Version 11.0 software to organize and classify data efficiently. The data will be analysed following a thematic analysis following the Braun & Clarke (2019) phases. First, three researchers independently will review all the transcriptions to gain familiarity with the data. Second, these researchers will select text fragments related to teachers' perceptions of the effects of the training program and subsequent implementation toward students. Finally, after the code review, the final themes and subthemes, containing the relevant meanings extracted from the dataset, will be further refined. It is expected that a deductive thematic analysis underpinned by the circumplex approach and SDT will be conducted because most of the questions are related to these frameworks. The other two researchers will supervise and share their viewpoints and interpretations to facilitate agreement during the data analysis process.

#### **Discussion**

One of the challenges faced by teachers and researchers is the difficulty of replicating interventions that have shown promising results. This endeavor is often hampered by inadequate reporting of intervention protocols and content. Providing a detailed description of the training program and the subsequent intervention may facilitate scalability to other areas, countries, and contexts. To fill this gap, the present study aims to comprehensively describe the protocol of a motivational training program, based on the circumplex model, aimed at

improving the autonomy-supportive and structuring teaching approaches and minimizing controlling and chaotic styles among PE teachers.

This study will provide a unique contribution to knowledge in ten key areas: (1) it will be the first motivational training program based on the recent circumplex model, due to the recent and innovative nature of this approach, and the eight teaching approaches proposed by the circumplex model will be assessed using real-life educational situations thought the SIS-PE instrument; (2) the quality of each face-to-face training session and follow-up sessions of the training program will be examined through short questionnaires at the end of each class, as well as a focus group with the entire PE teachers; (3) the effects of the intervention on a wide range of study variables will be evaluated using a mixed-method approach (i.e., questionnaires and focus groups) in both teachers and students; (4) the effects of the intervention on boys and girls students and male and female teachers will be examined; (5) not only a post-test, but also an intermediate measure will be used to examine how the study variables vary throughout the program; (6) the training program will not only take place before the implementation of the intervention, but also during the intervention; (7) the training program will include two individual and group follow-up sessions in which constructive feedback will be provided, as well as an individualized report; (8) promising strategies that have been shown to be effective in previous SDT-training programs (e.g., congruent style, brief theoretical part, real videos of PE teachers, microteaching, co-creation of teaching strategies, etc.) will be used; (9) the assessment of intervention fidelity through a new validated observational instrument in line with the circumplex model (i.e., SIS-PE-Coder) will be used; (10) MBCTs provided by Ahmadi et al. (2023) will be used in the development of the intervention implementation to find out to which behaviour change techniques are attributed to the intervention effects.

Likewise, some of the expected results for both teachers and students about the development of this training program will be presented according to the three hypotheses. Regarding the first hypothesis, as promising strategies used in previous SDT-training programs will be used (e.g., Aelterman et al., 2013), experimental group teachers will positively perceive the training program (e.g., innovation, practical usefulness, feasibility of the motivating strategies, intention to implement the motivating strategies, satisfaction, etc.). Teachers' feedback will help to make changes to the training program before it is disseminated to other areas, countries or contexts. This could enhance the acceptability, sustainability, and scalability of the training program.

Concerning the second hypothesis, experimental school female and male teachers are expected to perceive improvements in several antecedents, autonomy and competence satisfaction/frustration at work, (de)motivating teaching styles/approaches, and (mal)adaptive outcomes at least at the end of the intervention implementation toward students. According to SDT, teachers are expected to improve malleable antecedents such as (de)motivating teaching style beliefs due to scientific evidence or viewing videos of real classrooms of PE teachers. According to SDT, the improvement of the different antecedents could, in turn, improve autonomy and competence satisfaction/frustration at work (Aelterman et al., 2016; Matosic et al., 2016). The larger repertoire of teaching strategies learned during the training program may also enhance teachers' autonomy and competence satisfaction at work, as well as reduce teachers' autonomy and competence frustration at work, as they feel they have more resources to cope with their teaching. Finally, according to previous studies in PE teachers, autonomy and competence satisfaction at work could favour greater job satisfaction and job performance (Abós et al., 2018), as well as greater use of autonomy-supportive (i.e., participative and attuning) and structuring styles (i.e., guiding and clarifying) (Burgueño, Abós, et al., 2024; García-Cazorla et al., 2024). Conversely, reduction of autonomy and

competence frustration at work could favour lower emotional exhaustion (Abós et al., 2018), as well as a lower use of controlling (i.e., demanding and domineering approaches) and chaotic styles (i.e., abandoning and awaiting approaches) toward students (Burgueño, Abós, et al., 2024; García-Cazorla et al., 2024).

Finally, regarding the third hypothesis, it is expected that both boys and girls from the experimental groups will perceive improvements in (de)motivating teaching styles/approaches because of the implementation of strategies by their PE teachers over approximately five months (Vasconcellos et al., 2020). According to SDT, when students perceive that their PE teachers use autonomy support and structure, they are likely to feel autonomy and competence satisfied. Conversely, if they perceive controlling and chaotic teaching styles, they are likely to feel autonomy and competence frustrated (Vasconcellos et al., 2020). Finally, it is expected that through the improvement of need-based experiences, students will achieve improvements in affective (i.e., PE experiences), cognitive (i.e., learning in PE), and behavioural (i.e., intention to be physically active) outcomes (Vasconcellos et al., 2020).

#### Limitations

Some of the limitations in the development of the teacher training program are as follows. Firstly, the training duration could be kept brief to ensure that PE teachers grasp and internalize the motivational strategies, enabling them to effectively integrate these techniques into their PE classes. Acquiring new knowledge necessitates dedicated time for learning and assimilation, as well as opportunities for practice and self-and co-assessment. Nevertheless, an excessively lengthy training program might risk discouraging participation from PE teachers. In the scientific literature, these programs typically range from three to 12 hours, but there is no consensus regarding the ideal duration. If all teachers express a willingness to continue the training program, the possibility of slightly increasing the number of hours can

be considered. Secondly, observation will be used twice to ensure intervention fidelity and provide constructive feedback to teachers during the intervention but will not be used as a complementary measure of students' and teachers' perception of (de)motivating teaching styles in the three measures of the study due to lack of human resources. Thirdly, teachers' perceptions of their beliefs regarding (de)motivating teaching styles will not be assessed by means of questionnaires due to their length, as well as the absence of validated instruments of control and chaos styles. Additionally, relatedness satisfaction and frustration at work will not be assessed because the training program will not target teachers within the same school. Additionally, teachers' perceptions of depersonalization and reduced personal accomplishment (i.e., burnout factors) will not be assessed using questionnaires due to their length. However, all these variables will be assessed through the focus groups to obtain more information on the effects of the training program and the subsequent intervention carried out. Finally, students' perceptions of relatedness satisfaction and frustration in PE will not be assessed employing questionnaires due to their length and because the teacher training program was based on the circumplex model, which does not address the need for relatedness. As a final limitation, it is very likely that a post-intervention follow-up measure cannot be carried out the following academic year because in Spain it is very common for teachers to change schools every year. Therefore, it will only be possible to assess students' perception of the study variables if the teacher is the same. Similarly, the perception of (de)motivating teaching style might change with different classroom groups.

### **Conclusions**

The present study presents a comprehensive overview of the protocol for a training program designed for in-service PE teachers, based on the circumplex model, to maximize transparency and replicability. It is hoped that the motivational training program will help PE teachers in supporting autonomy and structure while minimizing the use of controlling and

chaotic teaching styles. This in turn may lead to an improvement in motivational-related variables and adaptive outcomes not only in students, but also in teachers. If the results are promising, this study can drive the professional development of motivational training programs for in-service PE teachers.

# **Funding statement**

This manuscript is part of the project "Assessing and improving teaching behaviors in Physical Education to improve students' motivational processes and Physical Activity levels (PE&PA project)" (PID2021-127897NA-I00) founded by MCIN /AEI /10.13039/501100011033 / FEDER, UE) and by "ERDF A way of making Europe". Javier García-Cazorla was specifically supported by a grant from the Government of Aragon.

## **Authors' contributions:**

Javier García-Cazorla<sup>1\*</sup>, Javier Sevil-Serrano<sup>2</sup>, Luis García González<sup>1</sup> and Ángel Abós<sup>1</sup> Faculty of Health and Sport Sciences. EFYPAF "Physical Education and Physical Activity Promotion"

Javier García-Cazorla https://orcid.org/0000-0001-8245-349X j.garcia@unizar.es

Luis García-González https://orcid.org/0000-0001-8115-0649 lgarciag@unizar.es

Sergio Diloy-Peña https://orcid.org/0000-0003-1357-9771 sdiloy@unizar.es

Rafael Burgueño https://orcid.org/0000-0003-2354-0037 rburgueno@uma.es

Ángel Abós https://orcid.org/0000-0002-1543-5109 aabosc@unizar.es

The authors report there are no competing interests to declare.

Research Group, University of Zaragoza, Huesca, Spain.

<sup>&</sup>lt;sup>2</sup> Faculty of Educational Science. Department of Education. University of Almeria, Andalucía, Spain.

<sup>\*</sup>Corresponding author: j.garcia@unizar.es

#### References

Abós, Á., Haerens, L., Sevil, J., Aelterman, N., & García-González, L. (2018). Teachers' motivation in relation to their psychological functioning and interpersonal style: A variable- and person-centered approach. *Teaching and Teacher Education*, 74, 21–34. https://doi.org/10.1016/j.tate.2018.04.010

- Abós, Á., Haerens, L., Sevil-Serrano, J., Morbée, S., Julián, J. A., & García-González, L. (2019). Does the level of motivation of physical education teachers matter in terms of job satisfaction and emotional exhaustion? A person-centered examination based on self-determination theory. *International Journal of Environmental Research and Public Health*, 16(16), 1–15. https://doi.org/10.3390/ijerph16162839
- Abós Catalán, Á., Sevil Serrano, J., Julián Clemente, J. A., Martín-Albo Lucas, J., & García-González, L. (2018). Spanish validation of the Basic Psychological Needs at Work Scale: A measure to predict teachers' well-being in the workplace. *International Journal for Educational and Vocational Guidance*, 18(2), 127–148.

  https://doi.org/10.1007/s10775-017-9351-4
- Aelterman, N., Vansteenkiste, M., Haerens, L., Soenens, B., Fontaine, J. R. J., & Reeve, J. (2019). Toward an integrative and fine-grained insight in motivating and demotivating teaching styles: The merits of a circumplex approach. *Journal of Educational Psychology*, 111(3), 497–521. https://doi.org/10.1037/edu0000293
- Aelterman, N., Vansteenkiste, M., Van Keer, H., De Meyer, J., Van den Berghe, L., & Haerens, L. (2013). Development and evaluation of a training on need-supportive teaching in physical education: Qualitative and quantitative findings. *Teaching and Teacher Education*, 29, 64–75. https://doi.org/10.1016/j.tate.2012.09.001
- Aelterman, N., Vansteenkiste, M., Van Keer, H., & Haerens, L. (2016). Changing teachers' beliefs regarding autonomy support and structure: The role of experienced psychological

- need satisfaction in teacher training. *Psychology of Sport and Exercise*, 23, 64–72. https://doi.org/10.1016/j.psychsport.2015.10.007
- Ahmadi, A., Noetel, M., Parker, P., Ryan, R. M., Ntoumanis, N., Reeve, J., Beauchamp, M.,
  Dicke, T., Yeung, A., Ahmadi, M., Bartholomew, K., Chiu, T. K. F., Curran, T., Erturan,
  G., Flunger, B., Frederick, C., Froiland, J. M., González-Cutre, D., Haerens, L., ...
  Lonsdale, C. (2023). A classification system for teachers' motivational behaviors
  recommended in self-determination theory interventions. *Journal of Educational Psychology*. https://doi.org/10.1037/edu0000783
- Barrick, M. R., Stewart, G. L., & Piotrowski, M. (2002). Personality and job performance:

  Test of the mediating effects of motivation among sales representatives. *Journal of Applied Psychology*, 87(1), 43–51. https://doi.org/10.1037/0021-9010.87.1.43
- Bouten, A., Haerens, L., Van Doren, N., Compernolle, S., & De Cocker, K. (2023). An online video annotation tool for optimizing secondary teachers' motivating style: Acceptability, usability, and feasibility. *Teaching and Teacher Education*, *134*, 104307. https://doi.org/10.1016/j.tate.2023.104307
- Braun, V., & Clarke, V. (2019). Reflecting on reflexive thematic analysis. *Qualitative Research in Sport, Exercise and Health*, 11(4), 589–597. https://doi.org/10.1080/2159676X.2019.1628806
- Burgueño, R., Abós, Á., Sevil-Serrano, J., Haerens, L., De Cocker, K., & García-González, L. (2024). A Circumplex Approach to (de)motivating Styles in Physical Education:

  Situations-In-School-Physical Education Questionnaire in Spanish Students, Pre-Service, and In-Service Teachers. *Measurement in Physical Education and Exercise Science*. https://doi.org/10.1080/1091367X.2023.2248098
- Burgueño, R., García-González, L., Abós, Á., & Sevil-Serrano, J. (2024). Students' motivational experiences across profiles of perceived need-supportive and need-

- thwarting teaching behaviors in physical education. *Physical Education and Sport Pedagogy*, 29(1), 82–96. https://doi.org/10.1080/17408989.2022.2028757
- Chen, B., Vansteenkiste, M., Beyers, W., Boone, L., Deci, E. L., Van der Kaap-Deeder, J.,
  Duriez, B., Lens, W., Matos, L., Mouratidis, A., Ryan, R. M., Sheldon, K. M., Soenens,
  B., Van Petegem, S., & Verstuyf, J. (2015). Basic psychological need satisfaction, need
  frustration, and need strength across four cultures. *Motivation and Emotion*, 39(2), 216–236. https://doi.org/10.1007/s11031-014-9450-1
- Cheon, S. H., & Reeve, J. (2015). A classroom-based intervention to help teachers decrease students' amotivation. *Contemporary Educational Psychology*, 40, 99–111. https://doi.org/10.1016/j.cedpsych.2014.06.004
- Cheon, S. H., Reeve, J., & Vansteenkiste, M. (2020). When teachers learn how to provide classroom structure in an autonomy-supportive way: Benefits to teachers and their students. *Teaching and Teacher Education*, *90*, 103004. https://doi.org/10.1016/j.tate.2019.103004
- Conesa, P. J., Duñabeitia, J. A., Onandia-Hinchado, I., & González-Cutre, D. (2023).

  Satisfying students' psychological needs in the classroom: Benefits of an online intervention to help primary school teachers during a pandemic academic year. *Teaching and Teacher Education*, 133, 104281. https://doi.org/10.1016/j.tate.2023.104281
- Diloy-Peña, S., Abós, Á., Sevil-Serrano, J., García-Cazorla, J., & García-González, L. (2024). Students' perceptions of physical education teachers' (de)motivating styles via the circumplex approach: Differences by gender, grade level, experiences, intention to be active, and learning. *European Physical Education Review*. https://doi.org/10.1177/1356336X241229353
- Escriva-Boulley, G., Guillet-Descas, E., Aelterman, N., Vansteenkiste, M., Van Doren, N., Lentillon-Kaestner, V., & Haerens, L. (2021). Adopting the situation in school

questionnaire to examine Physical Education teachers' motivating and demotivating styles using a circumplex approach. *International Journal of Environmental Research and Public Health*, *18*(14), 7342. https://doi.org/10.3390/ijerph18147342

- Field, A. (2017). *Discovering statistics using IBM SPSS statistics* (5th ed.). SAGE Publications.
- García-Cazorla, J., García-González, L., Burgueño, R., Diloy-Peña, S., & Abós, Á. (2024).

  What factors are associated with physical education teachers' (de) motivating teaching style? A circumplex approach. https://doi.org/10.1177/1356336X241248262
- Gil-Monte, P. R. (2002). *Validez factorial de la adaptación al español del Maslach Burnout Inventory-General Survey*. http://www.insp.mx/salud/index.html
- González, S. T., López, M. C. N., Marcos, Y. Q., & Rodríguez-Marín, J. (2012). Development and Validation of the Theory of Planned Behavior Questionnaire in Physical Activity. *The Spanish Journal of Psychology*, 15(2), 801–816.

  https://doi.org/10.5209/rev\_SJOP.2012.v15.n2.38892
- Haerens, L., Vansteenkiste, M., Aelterman, N., & Van den Berghe, L. (2016). Toward a
  Systematic Study of the Dark Side of Student Motivation: Antecedents and
  Consequences of Teachers' Controlling Behaviors. In *Building Autonomous Learners*(pp. 59–81). Springer Singapore. https://doi.org/10.1007/978-981-287-630-0
- Hedges, L. V., & Hedberg, E. C. (2007). Intraclass Correlation Values for Planning Group-Randomized Trials in Education. *Educational Evaluation and Policy Analysis*, 29(1), 60–87. https://doi.org/10.3102/0162373707299706
- Jang, H.-R., Cheon, S. H., Reeve, J., Song, Y.-G., & Lee, Y. (2023). Two ways teachers can develop greater harmonious passion. *Physical Education and Sport Pedagogy*, 1–16. https://doi.org/10.1080/17408989.2023.2206832

Matosic, D., Ntoumanis, N., & Quested, E. (2016). Antecedents of Need Supportive and Controlling Interpersonal Styles From a Self-Determination Theory Perspective: A Review and Implications for Sport Psychology Research. In *Sport and Exercise Psychology Research* (pp. 145–180). Elsevier. https://doi.org/10.1016/B978-0-12-803634-1.00007-8

- McConnell, M. M., Monteiro, S., & Bryson, G. L. (2019). Sample size calculations for educational interventions: principles and methods. In *Canadian Journal of Anesthesia* (Vol. 66, Issue 8, pp. 864–873). Springer New York LLC. https://doi.org/10.1007/s12630-019-01405-9
- Meerits, P. R., Tilga, H., & Koka, A. (2022). Fostering Need-Supportive Behaviors in Physical Education Teachers and Parents: A Cluster Randomized Controlled Trial Study Protocol of a Web-Based Intervention on Secondary School Students' Physical Activity. Methods and Protocols, 5(5). https://doi.org/10.3390/mps5050083
- Richards, K. A., Washburn, N. S., & Hemphill, M. A. (2019). Exploring the influence of perceived mattering, role stress, and emotional exhaustion on physical education teacher/coach job satisfaction. *European Physical Education Review*, *25*(2), 389–408. https://doi.org/10.1177/1356336X17741402
- Reeve, J., & Cheon, S. H. (2021). Autonomy-supportive teaching: Its malleability, benefits, and potential to improve educational practice. *Educational Psychologist*, *56*(1), 54–77. https://doi.org/10.1080/00461520.2020.1862657
- Reeve, J., Ryan, R. M., Cheon, S. H., Matos, L., & Kaplan, H. (2022). Supporting Students'

  Motivation. Routledge. https://doi.org/10.4324/9781003091738
- Reeve, J., Vansteenkiste, M., Assor, A. *et al.* The beliefs that underlie autonomy-supportive and controlling teaching: A multinational investigation. *Motiv Emot* 38, 93–110 (2014). https://doi.org/10.1007/s11031-013-9367-0

Ryan, R. M., & Deci, E. L. (2017). Self-determination theory: Basic psychological needs in motivation, development, and wellness. Guilford Publishing. https://doi.org/10.1521/978.14625/28806

- Skaalvik, E. M., & Skaalvik, S. (2011). Teacher job satisfaction and motivation to leave the teaching profession: Relations with school context, feeling of belonging, and emotional exhaustion. *Teaching and Teacher Education*, 27(6), 1029–1038. https://doi.org/10.1016/j.tate.2011.04.001
- Slemp, G. R., Field, J. G., & Cho, A. S. H. (2020). A meta-analysis of autonomous and controlled forms of teacher motivation. *Journal of Vocational Behavior*, *121*, 103459. https://doi.org/10.1016/j.jvb.2020.103459
- Slingerland, M., Borghouts, L., Jans, L., Weeldenburg, G., van Dokkum, G., Vos, S., & Haerens, L. (2017). Development and optimisation of an in-service teacher training programme on motivational assessment in physical education. *European Physical Education Review*, 23(1), 91–109. https://doi.org/10.1177/1356336X16639212
- Van Doren, N., De Cocker, K., Flamant, N., Compernolle, S., Vanderlinde, R., & Haerens, L. (2023). Observing physical education teachers' need-supportive and need-thwarting styles using a circumplex approach: how does it relate to student outcomes? *Physical Education and Sport Pedagogy*, 1–25. https://doi.org/10.1080/17408989.2023.2230256
- Vansteenkiste, M., Aelterman, N., Haerens, L., & Soenens, B. (2019). Seeking Stability in Stormy Educational Times: A Need-based Perspective on (De)motivating Teaching Grounded in Self-determination Theory. In *Advances in Motivation and Achievement* (Vol. 20, pp. 53–80). https://doi.org/10.1108/S0749-742320190000020004
- Vansteenkiste, M., Ryan, R. M., & Soenens, B. (2020). Basic psychological need theory:

  Advancements, critical themes, and future directions. *Motivation and Emotion*, 44(1), 1–31. https://doi.org/10.1007/s11031-019-09818-1

Vasconcellos, D., Parker, P. D., Hilland, T., Cinelli, R., Owen, K. B., Kapsal, N., Lee, J., Antczak, D., Ntoumanis, N., Ryan, R. M., & Lonsdale, C. (2020). Self-determination theory applied to physical education: A systematic review and meta-analysis. *Journal of Educational Psychology*, 112(7), 1444–1469. https://doi.org/10.1037/edu0000420

- White, R. L., Bennie, A., Vasconcellos, D., Cinelli, R., Hilland, T., Owen, K. B., & Lonsdale,
  C. (2021). Self-determination theory in physical education: A systematic review of
  qualitative studies. *Teaching and Teacher Education*, 99, 103247.
  https://doi.org/10.1016/j.tate.2020.103247
- Zamarripa, J., Rodríguez-Medellín, R., Pérez-Garcia, J. A., Otero-Saborido, F., & Delgado, M. (2020). Mexican Basic Psychological Need Satisfaction and Frustration Scale in Physical Education. *Frontiers in Psychology*, 11.
  https://doi.org/10.3389/fpsyg.2020.00253